CLINICAL TRIAL: NCT02883712
Title: Study of Predictors of Response to Anti Epilepsy in Epilepsy
Acronym: RESISTANT
Status: Terminated | Type: Observational
Why Stopped: defect inclusion
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2011_37; 2012-A00916-37 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-08-16; First posted 2016-08-30 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Seizure
Keywords: epilepsy; pharmacoresistant; antiepileptic drug; pharmacokinetic; pharmacodynamic; pharmacogenetic
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasmatic and serum samples for the dosage of the drugs Leucocytes for the intracellular dosage of the drugs DNA for pharmacogenetics analysis of the metabolism and pharmacodynamic targets of the drugs DNA for the genetic causes of epilepsy
Oversight: Data Monitoring Committee: No

SUMMARY:
Pharmacoresistant epilepsy remains around 30% despite the development of 25 anti epileptic drugs. Of course, this can be explained by pharmacoresistant epileptic brain diseases, as exemplified by some genetic diseases. However, the lack of specific guidelines for the choice of the anti epileptic drugs (apart from generalized and partial epilepsy) and the very large number of drugs with different and sometimes complex metabolism are challenges for neurologists. Among the 30 % of pharmacoresistant epilepsy, there is a part related to pharmacokinetic drawbacks that could be overcome with a more rigorous approach (i.e. dosage and pharmacogenetics tools). Moreover, the new anti epileptic drugs have metabolism more unrelated with the cytochrome P450 and less generalised adverse events. However, their metabolism could be more complexe (i.e. the less known Uridine 5'-diphospho-glucuronyltransferase (UGT) pathway) and bring more insidious neurological adverse events (i.e. depression, anxiety exacerbation, cognitive disorders worsening) which could largely impede the observance and the quality of life even if the number of seizure is reduced or not. The goal is to determine the predictive and the modulating factors of pharmacoresistance with a global analysis (i.e. whatever the anti epileptic drugs) and with a specific analysis (drug by drug) from a cohort of 1000 patients.

DETAILED DESCRIPTION:
The goal is to determine the predictive and the modulating factors of pharmacoresistance with a global analysis (i.e. whatever the anti epileptic drugs) and with a specific analysis (drug by drug with their specific metabolism pathways) from a cohort of 1000 patients. The response to the antiepileptic drugs modification will be analyse 3 months after the modification, with the analysis of the number of seizures, the quality of life, the Clinical Global Impression, the adverse events, the systematic dosage of all the molecules (residual concentration just before the taken) and the pharmacogenetic analysis of the main metabolism pathways and the main pharmacodynamic targets.

ELIGIBILITY:
Inclusion Criteria:

* Epileptic patients who required a treatment adaptation

Exclusion Criteria:

* patients unable to give reliable information and without caregiver
* pregnancy
* Severe comorbidity, which would impede interpretation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to our center with epilepsy (pharmacoresistant or pharmacosensitive)
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2013-05-21 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Clinical global impression of the patient | 3 months
  Clinical global impression assessment

SECONDARY OUTCOMES:
Number of seizure | 3 months
  recorded on the agenda of patients
Quality of life | 3 months
  Analyse with the Quality Of Life In Epilepsy Questionnaire
Adverse events | 3 months
  reported by the patients with a particular attention to attention and concentration worsening on interview
Concentration of the anti epileptic drug | 3 months
  plasmatic drug concentration will be systematically
Pharmacogenetics of the uridine 5'-diphosphate glucuronosyltransférases (UGT1A1, UGT2B7, UGT1A4) | 3 months
  the metabolism pathways of the drug
Pharmacogenetics of the Cytochrome P450 (2D6, 2C9, 2C19) | 3 months
  the metabolism pathways of the drug
Depression inventory for epilepsy | 3 months
  Neurological Disorders Depression Inventory for Epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: David DEVOS, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No